CLINICAL TRIAL: NCT01272388
Title: Aortic Stenosis and PhosphodiEsterase iNhibition With Aortic Valve Replacement (ASPEN-AVR): A Pilot Study
Acronym: ASPEN-AVR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: We designed a different pilot trial based on data obtained after this study started - the 2 studies were too overlapping to continue both.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Brian Lindman, MD, Assistant Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-1334a
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Aortic Stenosis
Keywords: Aortic valve stenosis; Tadalafil; Phosphodiesterase inhibitors; Hypertension, pulmonary; Hypertrophy, left ventricular
MeSH Terms: conditions — Aortic Valve Stenosis; Hypertension, Pulmonary; Hypertrophy, Left Ventricular | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tadalafil (Active Comparator)
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — Active drug will be encapsulated to look identical to the placebo pill. Subjects will take a single oral dose of tadalafil once daily from the time of randomization until the surgical date (~4 weeks). Subjects will begin by taking 20 mg (1 pill) daily for 3 days before having the dose increased to 40 mg (2 pills) once daily. If the increase to 40mg daily is not tolerated, then the dose will be decreased back to 20mg daily.
  Other Names: Cialis; Adcirca
  Arms: Tadalafil
Drug: Placebo — The placebo pill will be encapsulated to look identical to the active drug pill. Subjects will take a single oral dose of placebo once daily from the time of randomization until the surgical date (~4 weeks). Subjects will begin by taking 1 pill daily for 3 days before having the dose increased to 2 pills once daily. If the increase to 2 pills daily is not tolerated, then the dose will be decreased back to 1 pill daily.
  Arms: Placebo

SUMMARY:
Currently, aortic stenosis (AS) is considered a "surgical disease" with no medical therapy available to improve any clinical outcomes, including symptoms, time to surgery, or long-term survival. Thus far, randomized studies involving statins have not been promising with respect to slowing progressive valve stenosis. Beyond the valve, two common consequences of aortic stenosis are hypertrophic remodeling of the left ventricle (LV) and pulmonary venous hypertension; each of these has been associated with worse heart failure symptoms, increased operative mortality, and worse long-term outcomes. Whether altering LV structural abnormalities, improving LV function, and/or reducing pulmonary artery pressures with medical therapy would improve clinical outcomes in patients with AS has not been tested. Animal models of pressure overload have demonstrated that PDE5 inhibition influences NO-cGMP signaling in the LV and favorably impacts LV structure and function, but this has not been tested in humans with AS. Studies in humans with left-sided heart failure and pulmonary venous hypertension have shown that PDE5 inhibition improves functional capacity and quality of life, but patients with AS were not included in those studies. The investigators hypothesize that PDE5 inhibition with tadalafil will upregulate NO-cGMP signaling, reduce oxidative stress, and have a favorable impact on LV structure and function as well as pulmonary artery pressures and quality of life. In this pilot study, the investigators anticipate that short-term administration of tadalafil to patients with AS will be safe and well-tolerated.

DETAILED DESCRIPTION:
Patients with severe symptomatic AS who will undergo elective aortic valve replacement will be eligible for this randomized, double-blind, placebo-controlled, pilot study. Prior to randomization, subjects will have testing including: 6 minute walk, quality of life questionnaire, blood draw, and an echocardiogram. If an initial monitored dose of tadalafil is tolerated, participants will be randomized 2:1 to tadalafil vs. placebo. After 4 weeks on drug or placebo, subjects will have the same baseline testing repeated. At the time of aortic valve replacement surgery, the aortic valve and a small piece of LV myocardium will be taken for several analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe aortic stenosis (AVA < 1.0 cm2)
* Left ventricular hypertrophy
* EF ≥ 45%
* NYHA functional class ≥ 2
* Ambulatory (able to perform a 6 minute walk test)
* Normal sinus rhythm
* 18 years of age and older
* Able and willing to comply with all the requirements for the study

Exclusion Criteria:

* Need for ongoing nitrate medications
* SBP < 110mmHg or MAP < 75mmHg
* Moderately severe or severe mitral regurgitation
* Moderately severe or severe aortic regurgitation
* Creatinine clearance < 30 mL/min
* Increased risk of priapism
* Retinal or optic nerve problems or unexplained visual disturbance
* If a subject requires ongoing use of an alpha antagonist typically used for benign prostatic hyperplasia (BPH) (prazosin, terazosin, doxazosin, or tamsulosin), SBP < 120 mmHg or MAP < 80 mmHg is excluded
* Need for ongoing use of a potent CYP3A inhibitor or inducer (ritonavir, ketoconazole, itraconazole, rifampin)
* Cirrhosis
* Pulmonary fibrosis
* Current or recent (≤ 30 days) acute coronary syndrome
* O2 sat < 90% on room air
* Females that are pregnant or believe they may be pregnant
* Any condition which the PI determines will place the subject at increased risk or is likely to yield unreliable data
* Unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian R. Lindman, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tadalafil | Placebo
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: We designed a different pilot trial based on data obtained after this study started - the 2 studies were too overlapping to continue both. So, we stopped this study after enrollment of only 1 subject.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 69 |  | 69
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life as Assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: KCCQ overall summary score is reported. Scale is 0-100 (higher value is better).
Time Frame: Baseline and 4 weeks
Population: We designed a different pilot trial based on data obtained after this study started - the 2 studies were too overlapping to continue both. We stopped this study after only 1 patient (assigned to tadalafil) was enrolled.
Measure: Number; unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 1 | 0
units on a scale
  Baseline | 87 |
  4 weeks | 81.25 |

2. Secondary Outcome: 6 Minute Walk Distance
Description: How far the subject walked in 6 minutes.
Time Frame: Baseline and 4 weeks
Population: We designed a different pilot trial based on data obtained after this study started - the 2 studies were too overlapping to continue both. We only enrolled one participant (assigned to tadalafil) into the study before stopping the study.
Measure: Number; unit: feet
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 1 | 0
feet
  Baseline | 1080 |
  4 weeks | 860 |

ADVERSE EVENTS:
Arm/Group | Tadalafil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tadalafil (N=1) | Placebo (N=0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 — Patient described back discomfort/achiness for several hours that subsided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes